CLINICAL TRIAL: NCT07383935
Title: The Effect of Stress Ball on Anxiety, Fear and Vital Signs in Patients With Gastrointestinal System Cancer
Brief Title: Stress Ball Use During Chemotherapy in Gastrointestinal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, EMRE ERKAL, The Effect of Stress Ball on Anxiety, Fear, and Vital Signs in Patients With Gastrointestinal System Cancer, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GIS-STRESSBALL-2026
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal System Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Ball Intervention (Experimental): Participants in this arm will receive routine chemotherapy care and will additionally perform stress ball squeezing for 15 minutes starting at the beginning of the chemotherapy session. Patients will be instructed to inhale while squeezing the ball and exhale while releasing it, focusing attention on the activity.
  Interventions: Behavioral: Stress Ball
- Routine Care Control (No Intervention): Participants in this arm will receive routine chemotherapy care during their chemotherapy session and will not perform any stress ball or additional relaxation intervention.

INTERVENTIONS:
Behavioral: Stress Ball — The intervention consists of guided stress ball squeezing during chemotherapy. A round, medium-firm, compressible stress ball approximately 5-6 cm in diameter will be provided to participants. Starting at the beginning of the chemotherapy session, participants will squeeze the stress ball continuously for 15 minutes. They will be instructed to inhale while squeezing the ball, exhale while releasing their grip, and focus their attention on the squeezing activity. Disposable gloves will be used to maintain hygiene during the intervention. No additional behavioral or pharmacological interventions will be applied.
  Arms: Stress Ball Intervention

SUMMARY:
This study will investigate whether using a stress ball during chemotherapy can reduce anxiety, fear, and changes in vital signs in patients with gastrointestinal system cancers.

Patients receiving chemotherapy for gastrointestinal cancers often experience anxiety and fear, which may affect their heart rate, blood pressure, and breathing. A stress ball is a simple, low-cost, and safe method that may help patients relax during treatment.

In this randomized controlled study, 60 patients receiving chemotherapy will be assigned to either a stress ball group or a routine care group. Patients in the stress ball group will squeeze a stress ball for 15 minutes during their chemotherapy session. Anxiety, fear levels, and vital signs will be measured before and after chemotherapy in both groups.

The results of this study may help determine whether stress ball use is an effective non-drug method to improve emotional well-being and physiological stability in patients undergoing chemotherapy.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental trial designed to evaluate the effects of stress ball use during chemotherapy on anxiety, fear, and vital signs in patients with gastrointestinal system cancers.

Participants will be adult patients diagnosed with gastrointestinal system cancers who are receiving chemotherapy at the Artvin State Hospital Chemotherapy Unit. Eligible patients who provide informed consent will be randomly assigned in a 1:1 ratio to either an experimental group (stress ball intervention) or a control group (routine care).

Patients in the experimental group will be instructed to squeeze a medium-firm stress ball for 15 minutes starting at the beginning of their chemotherapy session. They will be guided to inhale while squeezing the ball and exhale while releasing it, focusing their attention on the activity. Patients in the control group will receive routine chemotherapy care without any additional intervention.

Anxiety and fear levels will be assessed before and after chemotherapy using validated measurement tools. Vital signs including blood pressure, heart rate, respiratory rate, body temperature, and oxygen saturation will also be recorded before and after the chemotherapy session. Outcomes will be compared between and within groups to determine the effectiveness of the stress ball intervention.

This study aims to provide evidence on whether a simple non-pharmacological method can improve psychological well-being and physiological stability during chemotherapy in patients with gastrointestinal system cancers.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 years or older
* Having a diagnosis of gastrointestinal system cancer and receiving chemotherapy
* Having no communication problems
* Having no physical disability that would prevent squeezing a stress ball
* Willingness to participate in the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-02-03 (Estimated)

PRIMARY OUTCOMES:
State Anxiety (STAI-State) score | Baseline (before chemotherapy session) and immediately after chemotherapy session

SECONDARY OUTCOMES:
Fear Severity (VAS-Fear) | Baseline (before chemotherapy session) and immediately after chemotherapy session
  Fear severity will be measured using a Visual Analog Scale (VAS-Fear). The change in scores before and after chemotherapy will be evaluated to assess the effect of the intervention on fear.
Systolic Blood Pressure | Baseline (immediately before chemotherapy session) and immediately after completion of the chemotherapy session.
  Systolic blood pressure measured using an automatic sphygmomanometer.
Diastolic Blood Pressure | Baseline (immediately before chemotherapy session) and immediately after completion of the chemotherapy session.
  Diastolic blood pressure measured using an automatic sphygmomanometer.
Heart Rate (Pulse) | Baseline (immediately before chemotherapy session) and immediately after completion of the chemotherapy session.
  Heart rate measured in beats per minute using an pulse oximeter
Respiratory Rate | Baseline (immediately before chemotherapy session) and immediately after completion of the chemotherapy session
  Respiratory rate measured by counting chest movements for one minute.
Body Temperature | Baseline (immediately before chemotherapy session) and immediately after completion of the chemotherapy session.
  Body temperature measured using a tympanic thermometer.
Oxygen Saturation (SpO₂) | Baseline (immediately before chemotherapy session) and immediately after completion of the chemotherapy session.

CONTACTS AND LOCATIONS:
Locations (1):
- Artvin State Hospital, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided